CLINICAL TRIAL: NCT00114062
Title: A Randomized, Double-Masked, Parallel Group, Multi-Center, Dose Ranging Pilot Study of Denufosol Tetrasodium (INS37217) Intravitreal Injection in Subjects With Uveitis Associated Macular Edema
Brief Title: Study to Treat Uveitis Associated Macular Edema
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06-103
Record Dates: First submitted 2005-06-13; First posted 2005-06-14 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Cystoid Macular Edema; Uveitis
Keywords: uveitis; macular edema; uveitis associated macular edema
MeSH Terms: conditions — Macular Edema; Uveitis | interventions — denufosol tetrasodium; Intravitreal Injections

INTERVENTIONS:
Drug: denufosol tetrasodium (INS37217) Intravitreal Injection

SUMMARY:
The purpose of this study is to determine whether denufosol tetrasodium (INS37217) Intravitreal Injection is well tolerated and has the potential to treat uveitis associated macular edema.

DETAILED DESCRIPTION:
Denufosol tetrasodium (INS37217) Intravitreal Injection may provide clinical benefit in treatment of uveitis associated macular edema (UME) by reducing retinal thickness as measured by OCT and possibly enabling recovery of vision loss associated with UME. Denufosol tetrasodium may also reverse the fluid accumulation of UME.

ELIGIBILITY:
Inclusion Criteria:

* Have anterior uveitis, intermediate uveitis, posterior uveitis or panuveitis in at least one eye
* Have persistent macular edema and uveitis whose conditions are stable
* Have no change in medication regimen for at least 3 months prior to randomization if currently taking medications such as immunosuppressive or anti-inflammatory agents; steroidal or non-steroidal agents (drops, oral or injected)
* Have an OCT scan with a qualifying retinal thickness in the study eye
* Have evidence of macular edema on OCT scan
* Have at lease one eligible eye to be treated in the study based on visual acuity.

Exclusion Criteria:

* Have proliferative vitreoretinopathy greater than grade B
* Have subretinal or vitreous hemorrhage, corneal opacity, or other conditions, which limit the view of the retina or obscure FA
* Have uncontrollable elevated IOP, advanced, previous filtration surgery, or any current evidence of endophthalmitis in the study eye
* Have ocular disorders in the study eye that may confound interpretation of study results
* Have had cataract surgery in the study eye within 3 months, YAG laser capsulotomy within the past 1 month, or any other intraocular surgery within the past 90 days
* Have pre-operative spherical equivalent refractive error of more than -10 diopters of myopia in the study eye
* Have had any intravitreal or periocular injection or corticosteroids in the study eye during the 3 months prior to screening
* Have any ocular implant device for the delivery of therapeutic agents to the eye
* Be taking any excluded medications that could obscure or confound study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2005-09; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of denufosol in subjects presenting with uveitis associated macular edema.
Assess the utility of denufosol in treating uveitis associated macular edema.

SECONDARY OUTCOMES:
Pilot study - not specified

CONTACTS AND LOCATIONS:
Overall Officials: Amy Schaberg, BSN, Study Director